CLINICAL TRIAL: NCT03610906
Title: Advancing Treatment for Pediatric Craniopharyngioma: Prospective Pilot Study Identifying Clinically Relevant Biological Targets for Medical Therapy
Brief Title: Prospective Pilot Study Identifying Clinically Relevant Biological Targets for Medical Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0426.cc
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Craniopharyngioma, Child
Keywords: Pilot Study; Biological Targets; CTNNB1; Tumor
MeSH Terms: conditions — Craniopharyngioma; Neoplasms | interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tissue and/or cyst fluid, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatrics with Tumors: Pediatrics who have a tumor specimen that is suspected to be craniopharyngioma, but is deemed superfluous to the clinical care of the patient (e.g. pathological diagnosis).
  Interventions: Procedure: Tumor and Blood Specimens

INTERVENTIONS:
Procedure: Tumor and Blood Specimens — If available, specimen will be sampled from within the tumor, and not include portions of the tumor capsule. If the tumor includes a cyst, fluid from the cyst will be sampled if available. For each tumor specimen, a companion sample of blood that would otherwise be disposed of through usual clinical practice in the operating room will also be collected.

SUMMARY:
New data suggests that the current treatment for pediatric adamantinomatous craniopharyngioma (CPA) may not be as effective as it could be.

DETAILED DESCRIPTION:
Current treatment regimens for pediatric CPA are limited to surgery and radiation therapy. This pilot study seeks to identify biologically rational therapeutics for the medical treatment of adamantinomatous CPA by confirming the overexpression of specific molecules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 0-21 years of age.
2. Patients with the diagnosis or clinical suspicion of craniopharyngioma in whom planned clinical management will include tissue sampling.

Exclusion Criteria:

1. Patients in whom final pathology does not demonstrate adamantinomatous craniopharyngioma
2. Patients in whom tissue specimen is not obtained/available
3. Patients over 21 years of age.
4. Patients who choose not to participate

Ages: 30 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population to be enrolled in this study will be children ages 0 through 21 years of age with a high preoperative suspicion of craniopharyngioma. The study population will be selected from the clinics at the 10 POETIC member institutions, and selected additional institutions by the treating clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2030-02-02 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of Potential Therapeutic Targets | Beginning of study to end of study, up to 1 year.
  Investigators will identify potential therapeutic targets through mRNA expression.
Identification of Potential Therapeutic Targets | Beginning of study to end of study, up to 1 year.
  Investigators will identify potential therapeutic targets through microarray analysis.
Identification of Potential Therapeutic Targets | Beginning of study to end of study, up to 1 year.
  Investigators will identify potential therapeutic targets immunohistochemistry.
Identification of Potential Therapeutic Targets | Beginning of study to end of study, up to 1 year.
  Investigators will identify potential therapeutic targets through quantitative PCR.
Identification of Potential Therapeutic Targets | Beginning of study to end of study, up to 1 year.
  Investigators will also perform immunostaining for beta-catenin and use DNA SNaPshot analysis to determine what parts of the tumor are responsible for observed gene signatures.

SECONDARY OUTCOMES:
Survival | Beginning of study up to age 21 or death, whichever comes first.
  The amount of time the patient survives with or without the disease.
Progression Free Survival (PFS) | Beginning of study up to age 21 or death, whichever comes first.
  The amount of time the patient survives without advancement of disease.
Visual Deficit Assessment | At 6 and 12 months after the specimen sample was taken.
  With regard to visual deficits, investigators will compare the rates of functional blindness, unilateral blindness, and visual field deficit.
Pituitary Function Assessment | At 6 and 12 months after the specimen sample was taken.
  With regard to pituitary function, investigators will assess patients based on the quality of life impairment that is associated with their dysfunction. Assessment will be divided among 4 groups:
  1. No dependence on hormone supplementation or evidence of diabetes insipidus
  2. Dependence on 1 or 2 hormone supplements without diabetes insipidus
  3. The presence of diabetes insipidus with or without the need for 2 or fewer hormone supplements
  4. Diabetes Insipidus with panhypopituitarism

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hankinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States